CLINICAL TRIAL: NCT03527446
Title: Sprint Interval Training: Insulin Sensitivity and Acute-Chronic Metabolic Flexibility in Individuals Living With Obesity: The i-FLEX Study
Brief Title: Acute and Chronic Metabolic Flexibility in Individuals Living With Obesity: The i-FLEX Study
Acronym: i-FLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Responsible Party: Principal Investigator, Martin Senechal, Assistant Professor, University of New Brunswick
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNewBrunswick
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Obesity; Endocrine; Insulin Sensitivity; Exercise
Keywords: Metabolic flexibility; Insulin sensitivity; Sprint interval training; Obesity; Exercise intensity
MeSH Terms: conditions — Obesity; Insulin Resistance; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Individuals living with obesity (BMI ≥ 30 km/m2; n=15) as well as normal weight (BMI ≥ 18.5 < 25.0 km/m2; n=15) adults (aged between 19 to 60 years) will be recruited to participate in the study. All participants will be asked to come in for a total of two visits and participate in a 4-week intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Weight (Experimental): BMI ≥ 18.5 < 25.0 km/m2 Sprint Interval Training
  Interventions: Behavioral: Sprint Interval Training
- Individuals living with Obesity (Experimental): BMI ≥ 30.0 km/m2 Sprint Interval Training
  Interventions: Behavioral: Sprint Interval Training

INTERVENTIONS:
Behavioral: Sprint Interval Training — The 4-week sprint interval intervention will consist of a work-rest ratio of four 30-s intervals of exercise at maximal capacity and 4-min of passive recovery at 50% of maximal capacity between intervals. There will be three sessions per week.

SUMMARY:
Regular exercise is a cornerstone in the prevention and the management of cardio-metabolic risk factors. Some of the beneficial effect of exercise training occurs through metabolic flexibility' enhancement. Metabolic flexibility is the ability to respond or adapt to conditional changes in metabolic demand, and previous literature has shown that individuals living with obesity have an impaired metabolic flexibility compared to lean individuals. However, there is a lack of empirical evidence on the impact of sprint interval training on metabolic flexibility and whether this translates into clinically meaningful outcomes.

This study will evaluate the impact of 4-week sprint interval training in normal weight individuals as well as individuals living with obesity on acute and chronic metabolic flexibility, irisin secretion and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Adults (Ages 19-60)
* Physically inactive for individuals living with obesity (not meeting Canadian Physical Activity Guidelines)
* Normal Weight (BMI ≥ 18.5 < 25.0 km/m2)
* Obesity (BMI ≥ 30.0 km/m2)

Exclusion Criteria:

* Individuals with Type 2 Diabetes.
* Individuals with impaired glucose tolerance.
* Individuals living with obesity that partake in regular exercise training / meet the Canadian Physical Activity Guidelines.
* Individuals with a condition or injury that may impact the ability to perform exercise or may be worsened by exercise.
* Individuals currently being treated with corticosteroids or atypical antipsychotics, as these agents significantly influence carbohydrate metabolism.
* have experienced >10% weight loss or enrolled in weight loss program within six months of enrolment.
* require use of medication(s) known to affect insulin sensitivity or secretion within the last 30 days.
* Medication(s) known to cause weight gain.
* weight loss medication(s).

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Metabolic Flexibility | Baseline and post-intervention (4 weeks)
  Chronic and acute metabolic flexibility will be quantified from the respiratory quotient (RQ) at rest and from the respiratory exchange ratio (RER) during a 4-6 minutes steady rate exercise bout.
Change in Insulin Sensitivity | Baseline and post-intervention (4 weeks)
  Insulin sensitivity will be measure with the Matsuda Index

SECONDARY OUTCOMES:
Change in Irisin | Baseline and post-intervention (4 weeks)
  This hormone will be quantified in the plasma during one acute session of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Senechal, PhD, Principal Investigator — University of New Brunswick
Locations (1):
- University of New Brunswick - Kinesiology, Fredericton, New Brunswick, Canada

REFERENCES:
- [Background] Muoio DM. Metabolic inflexibility: when mitochondrial indecision leads to metabolic gridlock. Cell. 2014 Dec 4;159(6):1253-62. doi: 10.1016/j.cell.2014.11.034. PMID 25480291